CLINICAL TRIAL: NCT02248532
Title: Repetitive Intramyocardial CD34+ Cell Therapy in Dilated Cardiomyopathy
Brief Title: Repetitive Intramyocardial CD34+ Cell Therapy in Dilated Cardiomyopathy (REMEDIUM)
Acronym: REMEDIUM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Bojan Vrtovec, Medical Director, Advanced Heart Failure and Transplantation, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REMEDIUM
Record Dates: First submitted 2014-09-16; First posted 2014-09-25 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Dilated Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): Repetitive stem cell administration
  Interventions: Biological: Stem cell therapy
- Group B (Active Comparator): Single stem cell administration
  Interventions: Biological: Stem cell therapy

INTERVENTIONS:
Biological: Stem cell therapy — Bone marrow cells will be mobilized into peripheral blood by daily subcutaneous injections of G-CSF (10 µg/kg daily) and collected by leukapheresis. Positive immunomagnetic selection of CD34+ cells will be performed. Electroanatomic mapping of the left ventricle will be performed using the Biosense NOGA system (Biosense-Webster®, Diamond Bar, CA). The target area for cell delivery will be defined as the myocardial segments with unipolar voltage potentials ≥8.3 mV, bipolar amplitudes >1.9 mV, and linear shortening <6%. Intramyocardial delivery of cell suspension will be performed with the MyoStar (BiosenseWebster®, Diamond Bar, CA) injection catheter. Each patient will receive 20 injections (0.3 mL each; total volume of 6 mL). All the procedures will be repeated 6 months after baseline.

SUMMARY:
The goal of REMEDIUM project is to develop personalized stem cell therapy for patients with chronic heart failure due to dilated cardiomyopathy (DCM). The main focus of the project is (1) on repetitive administration of cell therapy that would allow for long-lasting improvements in heart function and outcome in this patient population. In parallel, the investigators aim to (2) develop a standardized patient-specific stem cell product that could be cryopreserved and stored in a stem cell bank for prolonged time periods, and used for therapeutic application when clinically indicated. By using a unique multimodality imaging platform, the goal of this project is also to (3) define standardized clinical criteria that would serve as a guideline for evaluation of the effects of stem cell therapy in future clinical trials and everyday clinical settings. Finally, to improve the clinical implementation of cell therapy,the investigators aim to (4) develop a stem cell delivery technique that could be used to treat both left and right and ventricular failure and could be implemented in a standardized fashion designed for a widespread clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* Diagnosis of DCM according to European Society of Cardiology position statement
* Left ventricular ejection fraction (LVEF) by echocardiography 20-40%,
* New York Heart Association (NYHA) functional class heart failure II or III for at least 3 months before referral.

Exclusion Criteria:

* Acute multi-organ failure
* History of any malignant disease within 5 years
* Diminished functional capacity due to non-cardiac co-morbidities (COPD, PAOD, morbid obesity)
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction | baseline and 1 year
  The echocardiography data will be recorded and analyzed at the end of the study by an independent echocardiographer who will be blinded to the patient's treatment status and the timing of the recordings. Left ventricular end-systolic volume and end-diastolic volume and LVEF will be estimated using the Simpson's biplane method and left ventricular end-systolic dimension and end-diastolic dimension will be measured in the parasternal long axis view. All echocardiographic measurements will be averaged for 5 cycles.. The change in left ventricular ejection fraction (LVEF) between randomization and 1 year thereafter will be assessed by 2D echocardiography.

SECONDARY OUTCOMES:
Changes in regional wall motion | baseline and 1 year
  Left ventricular segmental wall motion analysis (strain) will be evaluated with TomTec software (TomTec Imaging Systems GmbH, Unterschleissheim, Germany), using a 17-segment model of the left ventricle.
Change in left ventricular dimension | 1 year
  The change in left ventricular dimensions between randomization and 1 year thereafter will be assessed by 2D echocardiography.
Change in exercise capacity | baseline and 1 year
  Change in exercise capacity will be evaluated by 6-minute walk test was performed by a blinded observer according to the standard protocol.
Change in NT-proBNP | baseline and 1 year

OTHER OUTCOMES:
Incidence of ventricular arrhythmias | 1 year
Cardiac mortality | 1 year
Hospitalization for heart failure | 1 year
Pump failure mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Please Select, Slovenia

REFERENCES:
- [Background] Vrtovec B, Poglajen G, Lezaic L, Sever M, Socan A, Domanovic D, Cernelc P, Torre-Amione G, Haddad F, Wu JC. Comparison of transendocardial and intracoronary CD34+ cell transplantation in patients with nonischemic dilated cardiomyopathy. Circulation. 2013 Sep 10;128(11 Suppl 1):S42-9. doi: 10.1161/CIRCULATIONAHA.112.000230. PMID 24030420
- [Derived] Vrtovec B, Poglajen G, Sever M, Zemljic G, Frljak S, Cerar A, Cukjati M, Jaklic M, Cernelc P, Haddad F, Wu JC. Effects of Repetitive Transendocardial CD34+ Cell Transplantation in Patients With Nonischemic Dilated Cardiomyopathy. Circ Res. 2018 Jul 20;123(3):389-396. doi: 10.1161/CIRCRESAHA.117.312170. Epub 2018 Jun 7. PMID 29880546
- [Derived] Frljak S, Jaklic M, Zemljic G, Cerar A, Poglajen G, Vrtovec B. CD34+ Cell Transplantation Improves Right Ventricular Function in Patients with Nonischemic Dilated Cardiomyopathy. Stem Cells Transl Med. 2018 Feb;7(2):168-172. doi: 10.1002/sctm.17-0197. PMID 29380563
- [Derived] Rozman JZ, Perme MP, Jez M, Malicev E, Krasna M, Novakovic S, Vrtovec B, Rozman P. The effect of CD34+ cell telomere length and hTERT expression on the outcome of autologous CD34+ cell transplantation in patients with chronic heart failure. Mech Ageing Dev. 2017 Sep;166:42-47. doi: 10.1016/j.mad.2017.06.001. Epub 2017 Jun 19. PMID 28636901